CLINICAL TRIAL: NCT04420598
Title: Multicenter, Open-Label, Single-Arm, Multicohort Phase II Clinical Trial of Trastuzumab Deruxtecan(DS-8201a) in Human Epidermal Growth Factor Receptor 2 HER2+ Advanced Breast Cancer With Brain Metastases and/or Leptomeningeal Carcinomatosis
Brief Title: DS-8201a for trEatment of aBc, BRain Mets, And Her2[+] Disease
Acronym: DEBBRAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDOPP243; 2019-001739-29 (EudraCT Number)
Record Dates: First submitted 2020-05-25; First posted 2020-06-09 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Advanced Breast Cancer; HER2-positive Breast Cancer; Brain Metastases; Leptomeningeal Metastasis
Keywords: Breast cancer; HER2; Brain metastases; Metastatic; unresectable; pretreated
MeSH Terms: conditions — Brain Neoplasms; Meningeal Carcinomatosis; Breast Neoplasms; Neoplasm Metastasis | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: This is a multicenter, international, open-label, single-arm, multicohort, two-stage optimal Simon's design, phase II clinical trial.
  After confirmed eligibility, patients will be assigned to one of the following five study cohorts:
  * Cohort 1: HER2-positive BC with non-progressing BM (after WBRT and/or SRS and or surgery.);
  * Cohort 2: HER2-positive or HER2-low BC with asymptomatic untreated BM;
  * Cohort 3: HER2-positive BC with progressing BMs after local treatment;
  * Cohort 4: HER2-low expressing BC with progressing BMs after local treatment;
  * Cohort 5: HER2-positive or HER2-low expressing BC with LMC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab deruxtecan (DS-8201a) (Experimental): * Cohort 1: HER2-positive BC with non-progressing BM (after WBRT and/or SRS and or surgery.);
  * Cohort 2: HER2-positive or HER2-low BC with asymptomatic untreated BM;
  * Cohort 3: HER2-positive BC with progressing BMs after local treatment;
  * Cohort 4: HER2-low expressing BC with progressing BMs after local treatment;
  * Cohort 5: HER2-positive or HER2-low expressing BC with LMC.
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — After having confirmed eligibility and entered into the clinical trial, patients will be treated with trastuzumab deruxtecan (DS-8201a) at 5.4 mg/Kg administered as an intravenous (IV) infusion on Day of 21-day cycle (Q3W), initially for at least 90 minutes, then, if there is no infusion-related reaction, for a minimum of 30 minutes.
  In patients with hormone receptor (HR)-positive status (estrogen receptor [ER] and/or progesterone receptor [PgR]) administration of endocrine therapy is not allowed.
  In patients allocated in study cohort 5, administration of intrathecal therapy is not allowed
  Other Names: (DS-8201a)

SUMMARY:
This is a multicenter, international, open-label, single-arm, multicohort, two-stage optimal Simon's design, phase II clinical trial

DETAILED DESCRIPTION:
Pretreated, unresectable locally advanced or metastatic Human Epidermal Growth Factor Receptor 2 (HER2)-positive or HER2-low expressing breast cancer (BC) with untreated or treated brain metastases (BMs) or leptomeningeal carcinomatosis (LMC).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF) prior to participation in any study-related activities.
2. Male or female patients ≥ 18 years at the time of signing ICF.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 for Cohorts 1 to 4 and 0-2 for cohort 5.
4. Life expectancy ≥ 12 weeks.
5. Histologically confirmed invasive breast cancer based on local testing on the most recent analyzed biopsy of the following breast cancer (BC) subtypes per 2018 American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) criteria:

   * Cohort 1 and 3: HER2 positive status
   * Cohort 4: HER2-low expressing status
   * Cohort 2 and 5: both HER2 positive and HER2-low expressing status

   Note 1: According to the 2018 ASCO-CAP guidelines, HER2- positive status is defined as HER2 immunohistochemistry (IHC) 3+, in situ hybridization (ISH) ≥ 2.0, or average HER2 copy number ≥ 6.0 signals. HER2-low expressing status defined as IHC 2+ / ISH-negative or IHC 1+ (ISH-negative or untested).

   Note 2: Central confirmation of HER2 is not required for study entry. However, tissue blocks, or slides, must be submitted to confirm BC subtype by a Sponsor-designated central laboratory retrospectively.
6. Unresectable locally advanced or metastatic disease documented by computerized tomography (CT) scan or magnetic resonance imaging (MRI) that is not amenable to resection with curative intent.
7. At least one brain lesion needed to be measurable (≥10 mm on T1-weighted, gadolinium-enhanced MRI) (study cohorts 2 to 4) or leptomeningeal carcinomatosis (LMC) with positive cerebrospinal fluid (CSF) cytology (study cohort 5).

   * Study cohort 1: History of BM that are non-progressing after WBRT and/or SRS and or surgery.
   * Study cohort 2: Presence of asymptomatic BM without clinical requirement for local intervention (WBRT and/or SRS and/or surgery).
   * Study cohorts 3 and 4: Evidence of new and/or progressive BM following previous WBRT and/or SRS and/or surgery.
   * Study cohort 5: Evidence of LMC with positive CSF cytology.
8. Previous treatments:

   * For HER2-positive patients have been previously treated with a taxane and at least one HER2-targeted therapy in the advanced scenario.
   * For HER2-low-expressing patients that also are endocrine receptor negative must have been previously treated with at least one chemotherapy regimen. If endocrine receptor positive, patients must have been previously treated with at least one chemotherapy and one endocrine regimen in the metastatic setting.
9. Patients must agree to collection of blood samples at the time of inclusion, at cycle 2 of treatment, and upon progression or study termination.

   Note: In study cohort 5: Patients must agree to perform spinal taps or must be willing to have an Ommaya reservoir placed for CSF assessment, at baseline, every three weeks for 12 weeks (corresponding to the first 5 cycles of treatment) and every six weeks thereafter.
10. Willingness and ability to provide tumor biopsy (if feasible) from metastatic lesions or breast primary tumor both at the time of the inclusion and after disease progression in order to perform exploratory studies.

    Note: If feasible, patients should provide a tissue sample at baseline from metastases amenable to biopsy (at sites of locoregional recurrence [skin, chest wall, breast or lymph nodes], or distant recurrence [bone, liver, lung or abdomen]) or as alternative from breast primary tumor, that will be obtained between progression to the prior regimen and inclusion in the study. Patients for whom tissue sample cannot be obtained (e.g., non-measurable disease, inaccessible tumor or subject safety concern) may submit an archived metastatic tumor specimen only upon agreement from the Sponsor. If feasible, an additional tissue sample should be collected at the end of treatment visit for patients who discontinue treatment due to disease progression.
11. Patients should have left ventricular ejection fraction (LVEF) ≥ 50% by either an echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before enrolment.
12. Adequate hematologic and organ function within 14 days before the first study treatment on Day 1 of Cycle 1, defined by the following:

    • Hematological: White blood cell (WBC) count 3 3.0 x 109/L, absolute neutrophil count (ANC) 3 1.5 x 109/L, platelet count 3 100.0 x109/L, and hemoglobin 3 9.0 g/dL. (Platelet, red blood cell transfusion as well as G-CSF administration are not allowed within 1 week of screening assessments).

    Hepatic: Bilirubin ≤ 1.5 times the upper limit of normal (× ULN) (< 3 x ULN in the case of documented Gilbert's disease and/or liver metastases); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 × ULN (in the case of liver metastases ≤ 5 × ULN); alkaline phosphatase (ALP) ≤ 2 × ULN (≤ 5 × ULN in the case of liver and/or bone metastases ≤ 5 × ULN), serum albumin 3 2.5 g/dL

    • Renal: Serum creatinine £ 1.5 × ULN or creatinine clearance ≥ 30 mL/min based on Cockcroft-Gault equation (*Cockcroft-Gault equation: ([{140 - age in years} × {ACTUAL WEIGHT in kg}] divided by [{72 × serum creatinine in mg/dL} multiplied by 0.85 if female])) Coagulation: International Normalized Ratio (INR)/Prothrombin Time (PT) and activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN (except for patients receiving anticoagulation therapy).

    Note: Patients receiving heparin treatment should have an aPTT) between 1.5 and 2.5 × ULN (or patient value before starting heparin treatment). Patients receiving coumarin derivatives should have an INR between 2.0 and 3.0 assessed in two consecutive measurements one to four days apart. Patients should be on a stable anticoagulant regimen.
13. Has adequate treatment washout period before enrollment, as indicated:

    1. Major surgery: > 4 weeks;
    2. Radiation therapy: > 4 weeks (palliative stereotactic radiation therapy to other areas ≥ 2 weeks);
    3. Anticancer systemic treatment (including immunotherapy, retinoid therapy, hormonal therapy): ≥ 3 weeks (≥ 2 weeks or 5 half-lives, whichever is longer, for small-molecule targeted agents such as 5-fluorouracil-based agents, folinate agents, weekly paclitaxel; ≥ 6 weeks for nitrosureas or mitomycin C);
    4. Antibody based anti-cancer therapy:≥ 4 weeks;
    5. Chloroquine/Hydroxychloroquine>14 days
14. Resolution of all acute toxic effects of prior anti-cancer therapy to grade ≤1 as determined by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5.0 (except for alopecia or other toxicities). Subjects with chronic Grade 2 toxicities may be eligible per the discretion of the Investigator after consultation with the Sponsor Medical Monitor or designee (e.g., Grade 2 chemotherapy-induced neuropathy).
15. Male and female subjects of reproductive/childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least 7 months for females and 4 months for males after the last dose of study drug. Methods considered as highly effective methods of contraception include:

    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

      i. Oral ii. Intravaginal iii. Transdermal
    * Progestogen-only hormonal contraception associated with inhibition of ovulation: iv. Oral v. Injectable vi. Implantable
    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion
    * Vasectomized partner
    * Complete sexual abstinence defined as refraining from heterosexual intercourse during and upon completion of the study and for at least 7 months after the last dose of study drug. Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not an acceptable method of contraception.

    Note: Non-child-bearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases, a blood sample with simultaneous follicle-stimulating hormone [FSH] > 40 mIU/mL and estradiol < 40 pg/mL [< 147 pmol/L] is confirmatory).
16. Male subjects must agree to not freeze or donate sperm starting at Screening and throughout the study period, and at least 7months after the final study drug administration. Preservation of sperm should be considered prior to enrolment in this study.
17. Female subjects must agree to not donate, or retrieve for their own use, ova from the time of Screening and throughout the study treatment period, and for at least 7 months after the final study drug administration.
18. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, post-treatment follow-up and other study procedures.

Exclusion Criteria:

Patients will be excluded from the study if they meet ANY of the following criteria:

1. Inability to comply with study and follow-up procedures.
2. Previous treatment with trastuzumab deruxtecan (DS-8201a) or any other antibody drug conjugate (ADC) which consists of an exatecan derivative that is a topoisomerase 1 inhibitor.
3. Medical history of myocardial infarction within 6 months before enrollment, symptomatic congestive heart failure (New York Heart Association Class II to IV), troponin levels consistent with myocardial infarction within 28 days prior to enrollment.
4. Corrected QT interval (QTc) prolongation to > 470 ms (females) or >450 ms (males) based on average of the screening triplicate12- lead ECG.
5. History of (non-infectious) interstitial lung disease (ILD) that required steroids, has current ILD, or where suspected ILD cannot be ruled out by imaging at screening.
6. Clinically significant corneal disease in the opinion of the Investigator.
7. Spinal cord compression.
8. Multiple primary malignancies within 3 years, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, other solid tumors curatively treated, or contralateral breast cancer.
9. History of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product.
10. History of severe hypersensitivity reactions to other monoclonal antibodies.
11. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
12. Patients with substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
13. Known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection. Subjects should be tested for HIV prior to enrollment if required by local regulations or institutional review board (IRB)/ethics committee (EC).
14. Female patients who are pregnant or breastfeeding or planning to become pregnant.
15. No other systemic therapy for metastatic disease including chemotherapy, immunotherapy, targeted therapy (small molecules/ monoclonal antibodies), or endocrine therapy
16. Major surgery (defined as requiring general anesthesia) or significant traumatic injury within 4 weeks of start of study drug, or patients who have not recovered from the side effects of any major surgery, or patients who may require major surgery during the study.
17. Radiotherapy within 4 weeks or limited-field palliative radiotherapy within 2 weeks prior to study enrolment, or patients who have not recovered from radiotherapy-related toxicities to baseline or grade ≤ 1 and/or from whom ≥ 25% of the bone marrow has been previously irradiated.
18. Use of concurrent investigational agents or other concomitant anticancer therapies.
19. Use of intrathecal therapy for LMC
20. Active bleeding diathesis, previous history of bleeding diathesis, or chronic anti-coagulation treatment (the use of low molecular weight heparin is allowed as soon as it is used as prophylaxis intention).
21. Serious concomitant systemic disorder (e.g., active infection including HIV, active hepatitis, liver cirrhosis, end stage chronic renal disease) incompatible with the study (at the discretion of investigator).
22. Any of the following within 6 months of enrollment: severe/unstable angina, ongoing cardiac dysrhythmias of NCI-CTCAE v.5.0 grade 32, coronary/peripheral artery bypass graft, cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
23. Uncontrolled electrolyte disorders of NCI-CTCAE v.5.0 grade ≥ 2.
24. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.), and any autoimmune, connective tissue or inflammatory disorders with potential pulmonary involvement (i.e. Rheumatoid arthritis, Sjogren's, sarcoidosis etc.), or prior pneumonectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Vaz Batista, MD, Principal Investigator — MedSIR
Locations (16):
- Portugal (2):
  - Champalimaud Center for the Unknown, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE (IPO Porto), Porto
- Spain (14):
  - Institut Català d'Oncologica ICO Badalona, Badalona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital del Mar, Barcelona
  - Institut Oncologic Baselga-Hospital Quiron Salud Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Institut Catala d'Oncologia ICO Hospitalet, L'Hospitalet de Llobregat
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - IOB- Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Fundación Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Migue Servet, Zaragoza

REFERENCES:
- [Derived] Vaz Batista M, Perez-Garcia JM, Garrigos L, Garcia-Saenz JA, Cortez P, Racca F, Blanch S, Ruiz-Borrego M, Fernandez-Ortega A, Fernandez-Abad M, Iranzo V, Gion M, Martrat G, Alcala-Lopez D, Perez-Escuredo J, Sampayo-Cordero M, Llombart-Cussac A, Braga S, Cortes J. The DEBBRAH trial: Trastuzumab deruxtecan in HER2-positive and HER2-low breast cancer patients with leptomeningeal carcinomatosis. Med. 2025 Jan 10;6(1):100502. doi: 10.1016/j.medj.2024.08.001. Epub 2024 Sep 11. PMID 39265579
- [Derived] Vaz Batista M, Perez-Garcia JM, Cortez P, Garrigos L, Fernandez-Abad M, Gion M, Martinez-Bueno A, Saavedra C, Teruel I, Fernandez-Ortega A, Servitja S, Ruiz-Borrego M, de la Haba-Rodriguez J, Martrat G, Perez-Escuredo J, Alcala-Lopez D, Sampayo-Cordero M, Braga S, Cortes J, Llombart-Cussac A. Trastuzumab deruxtecan in patients with previously treated HER2-low advanced breast cancer and active brain metastases: the DEBBRAH trial. ESMO Open. 2024 Sep;9(9):103699. doi: 10.1016/j.esmoop.2024.103699. Epub 2024 Sep 9. PMID 39255534

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: •Cohort 1: HER2-positive BC with non-progressing BM (after WBRT and/or SRS and or surgery.);
- Cohort 2: • Cohort 2: HER2-positive or HER2-low BC with asymptomatic untreated BM;
- Cohort 3: • Cohort 3: HER2-positive BC with progressing BMs after local treatment;
- Cohort 4: • Cohort 4: HER2-low expressing BC with progressing BMs after local treatment;
- Cohort 5: • Cohort 5: HER2-positive or HER2-low expressing BC with LMC.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 8 | 10 | 9 | 6 | 7
Completed | 3 | 3 | 1 | 4 | 2
Not Completed | 5 | 7 | 8 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 8 | 10 | 9 | 6 | 7 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (10.4) | 53.4 (13.5) | 50.2 (8.8) | 61.0 (9.5) | 52.7 (9.9) | 52.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 9 | 6 | 7 | 40
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ECOG [Count of Participants; unit: Participants] — The ECOG performance status evaluates participants' physical functioning, with lower values indicating better outcomes and higher values indicating worse physical impairment
  Participants
    0 | 5 | 9 | 6 | 1 | 3 | 24
    1 | 3 | 1 | 3 | 5 | 2 | 14
    2 | 0 | 0 | 0 | 0 | 2 | 2
Measurable disease at screening [Count of Participants; unit: Participants]
  No | 3 | 0 | 0 | 0 | 4 | 7
  Yes | 5 | 10 | 9 | 6 | 3 | 33
Number of metastatic organ sites [Count of Participants; unit: Participants]
  1 | 4 | 0 | 2 | 0 | 1 | 7
  2 | 1 | 2 | 5 | 0 | 5 | 13
  3 | 2 | 4 | 1 | 2 | 0 | 9
  4 | 0 | 2 | 1 | 1 | 0 | 4
  5 | 1 | 0 | 0 | 2 | 1 | 4
  6 | 0 | 2 | 0 | 0 | 0 | 2
  7 | 0 | 0 | 0 | 1 | 0 | 1
HER2 IHC test [Count of Participants; unit: Participants] — The HER2 IHC test evaluates HER2 protein expression in tumor cells on a 0 to 3+ scale:
  0: No staining or faint in <10% of cells.
  1. : Weak, incomplete staining in >10%.
  2. : Moderate, complete staining in >10%.
  3. : Strong, complete staining in >10%.
  Participants
    0 | 0 | 0 | 0 | 0 | 0 | 0
    1+ | 0 | 5 | 0 | 5 | 4 | 14
    2+ | 2 | 1 | 2 | 1 | 0 | 6
    3+ | 6 | 4 | 7 | 0 | 3 | 20
HER2 status [Count of Participants; unit: Participants]
  Positive | 8 | 4 | 9 | 0 | 3 | 24
  Low expressing | 0 | 6 | 0 | 6 | 4 | 16
  Negative | 0 | 0 | 0 | 0 | 0 | 0
  Indeterminate | 0 | 0 | 0 | 0 | 0 | 0
Estrogen receptor status [Count of Participants; unit: Participants]
  Negative | 4 | 3 | 2 | 3 | 2 | 14
  Positive | 4 | 7 | 7 | 3 | 5 | 26
Progesterone receptor status [Count of Participants; unit: Participants]
  Negative | 2 | 4 | 2 | 3 | 2 | 13
  Positive | 6 | 6 | 7 | 3 | 5 | 27
Hormone receptor status [Count of Participants; unit: Participants]
  Negative | 1 | 3 | 2 | 2 | 2 | 10
  Positive | 7 | 7 | 7 | 4 | 5 | 30
Number of previous early disease treatment lines [Count of Participants; unit: Participants]
  0 | 2 | 4 | 3 | 1 | 0 | 10
  1 | 0 | 2 | 2 | 2 | 0 | 6
  2 | 1 | 2 | 0 | 3 | 2 | 8
  3 | 3 | 1 | 3 | 0 | 4 | 11
  4 | 0 | 0 | 1 | 0 | 0 | 1
  5 | 1 | 0 | 0 | 0 | 1 | 2
  6 | 1 | 1 | 0 | 0 | 0 | 2
Number of previous early disease treatment lines [Mean (Standard Deviation); unit: Number of previous early disease treatm] | 2.8 (2.1) | 1.5 (1.9) | 1.7 (1.6) | 1.3 (0.8) | 3.0 (1.0) | 2.0 (1.7)
Previous early disease treatment line [Count of Participants; unit: Participants]
  No | 2 | 4 | 3 | 1 | 0 | 10
  Yes | 6 | 6 | 6 | 5 | 7 | 30
Previous early disease treatment [Count of Participants; unit: Participants]
  Antineoplastic agents | 6 | 5 | 6 | 5 | 7 | 29
  Endocrine therapy | 3 | 4 | 5 | 0 | 4 | 16
  Therapeutic radiopharmaceuticals | 3 | 2 | 3 | 1 | 2 | 11
  Immunosuppressants | 0 | 0 | 1 | 2 | 0 | 3
Previous lines in advanced disease [Count of Participants; unit: Participants]
  1 | 2 | 0 | 1 | 0 | 1 | 4
  2 | 2 | 1 | 3 | 1 | 1 | 8
  3 | 1 | 1 | 0 | 3 | 0 | 5
  4 | 1 | 2 | 0 | 2 | 2 | 7
  5 | 1 | 0 | 3 | 0 | 1 | 5
  6 | 0 | 1 | 0 | 0 | 1 | 2
  7 | 0 | 4 | 0 | 0 | 0 | 4
  8 | 1 | 1 | 0 | 0 | 1 | 3
  9 | 0 | 0 | 0 | 0 | 0 | 0
  10 | 0 | 0 | 0 | 0 | 0 | 0
  11 | 0 | 0 | 1 | 0 | 0 | 1
  12 | 0 | 0 | 0 | 0 | 0 | 0
  13 | 0 | 0 | 1 | 0 | 0 | 1
Previous advanced/ metastatic disease systemic treatment lines [Count of Participants; unit: Participants] | 8 | 10 | 9 | 6 | 7 | 40
Previous systematic cancer therapy [Count of Participants; unit: Participants]
  Trastuzumab | 7 | 3 | 9 | 1 | 3 | 23
  Trastuzumab emtansine | 4 | 2 | 6 | 0 | 3 | 15
  Pertuzumab | 7 | 3 | 5 | 0 | 3 | 18
  Other anti-HER2 therapy | 3 | 1 | 7 | 0 | 1 | 12
  Endocrine therapy | 3 | 7 | 4 | 4 | 3 | 21
  LHRH agonist therapy | 1 | 4 | 1 | 1 | 0 | 7
Previous systematic cancer therapy [Count of Participants; unit: Participants]
  Complete or partial response | 2 | 2 | 5 | 1 | 0 | 10
  Stable disease | 2 | 3 | 2 | 1 | 0 | 8
  Disease progression | 2 | 5 | 2 | 4 | 6 | 19
  Could not be elevated | 2 | 0 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: 16 Weeks PFS Per Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) (Cohort 1)
Description: This outcome measure evaluates progression-free survival (PFS) in Cohort 1 over a 16-week period, using the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria.
Time Frame: From baseline up to 16 weeks
Population: This outcome measure was the primary endpoint evaluated exclusively in Cohort 1. Therefore, results are only reported for the participants in this cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: HER2-positive BC with non-progressing BM (after WBRT and/or SRS and or surgery.);
Arm/Group | Cohort 1
Number analyzed (Participants) | 8
Participants
  With PFS at 16 weeks | 1
  Without PFS at 16 weeks | 7

2. Primary Outcome: Objective Response Rate According RANO-BM (Cohorts 2, 3 and 4)
Description: The proportion of patients achieving either Complete Response (CR) or Partial Response (PR) at any assessment time point, based on Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria
Time Frame: Each participant was assessed from baseline until the last tumor response evaluation, up to 16 months.
Population: This outcome measure was assessed only in Cohorts 2, 3, and 4. Therefore, data for Cohorts 1 and 5 are not included in this measure
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: HER2-positive or HER2-low BC with asymptomatic untreated BM;
- Cohort 3: HER2-positive BC with progressing BMs after local treatment;
- Cohort 4: HER2-low expressing BC with progressing BMs after local treatment;
Arm/Group | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 9 | 6
Participants
  No | 3 | 4 | 3
  Yes | 7 | 5 | 3

3. Primary Outcome: Overall Survival in Cohort 5
Description: Median of OS rate for patients
Time Frame: Each participant was assessed from baseline until the last tumor response evaluation, up to 16 months.
Population: Overall survival the primary outcome measure only in Cohort 5. Therefore, data for other cohorts are not included in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 5
Number analyzed (Participants) | 7
months | 13.3 [2.5 to NA] — Not enough events occurred after the median to calculate the top interval

4. Secondary Outcome: Intra-cranial Evaluation According to RANO-BM
Description: Each participant was assessed from baseline until the last tumor response evaluation, up to 16 months.
Time Frame: Each participant was assessed from baseline until the last tumor response evaluation, up to 16 months.
Population: Patients that have at least one CNS lesion
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 4 | 10 | 9 | 6 | 5
Participants
  CR | 2 | 0 | 0 | 0 | 1
  PR | 0 | 7 | 5 | 3 | 0
  SD≥24w | 2 | 1 | 1 | 1 | 3
  SD<24w | 0 | 2 | 2 | 2 | 1
  PD | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Extra-cranial Evaluation According to RECIST v1.1
Description: This outcome measure assesses the extra-cranial response of metastatic lesions outside the brain using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines.
Time Frame: Each participant was assessed from baseline until the last tumor response evaluation, up to 16 months.
Population: Patients that had at least one non-CNS lesion
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 7 | 10 | 5 | 6 | 6
Participants
  PR | 4 | 3 | 2 | 3 | 0
  CR | 0 | 0 | 0 | 0 | 0
  SD ≥24 weeks | 2 | 3 | 3 | 0 | 5
  SD <24 weeks | 0 | 3 | 0 | 3 | 0
  PD | 1 | 1 | 0 | 0 | 1

6. Secondary Outcome: Global Evaluation According to RECIST v1.1
Description: The global evaluation of tumor response will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. This includes classification into categories such as Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD), based on changes in tumor size and the appearance of new lesions.
Time Frame: Each participant was assessed from baseline until the last tumor response evaluation, up to 16 months.
Population: Patients with at least one CNS and non-CNS lesion
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 8 | 10 | 9 | 6 | 7
Participants
  PR | 4 | 3 | 2 | 2 | 0
  CR | 0 | 0 | 0 | 0 | 0
  SD ≥24 | 3 | 3 | 4 | 1 | 5
  SD <24 | 0 | 3 | 2 | 3 | 1
  PD | 1 | 1 | 1 | 0 | 1

7. Secondary Outcome: Unconfirmed Clinical Benefit Rate According to RANO-BM and RECIST v1.1
Description: The Clinical Benefit Rate (CBR) is a measure of the proportion of patients who achieve a clinically meaningful benefit from the treatment
Time Frame: Each participant was assessed from baseline until the last tumor response evaluation, up to 16 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 8 | 10 | 9 | 6 | 7
Participants
  No | 1 | 4 | 3 | 3 | 2
  Yes | 7 | 6 | 6 | 3 | 5

ADVERSE EVENTS:
Time Frame: Each participant was assessed from baseline until the last tumor response evaluation, up to 16 months.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 4/8 | 5/10 | 6/9 | 2/6 | 5/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/10 | 5/9 | 1/6 | 4/7
Other Adverse Events (participants affected / at risk) | 8/8 | 10/10 | 8/9 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=10) | Cohort 3 (N=9) | Cohort 4 (N=6) | Cohort 5 (N=7)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superinfection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=10) | Cohort 3 (N=9) | Cohort 4 (N=6) | Cohort 5 (N=7)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 4 (5) | 1 (1) | 1 (1) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (6) | 4 (6) | 2 (2) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 5 (8) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 3 (4) | 1 (2) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (9) | 3 (4) | 2 (3) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 4 (5) | 3 (6) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram QRS complex prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (11) | 9 (24) | 4 (10) | 5 (6) | 3 (4)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 3 (4) | 1 (3) | 2 (2) | 2 (5)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (6) | 3 (3) | 2 (2) | 0 (0) | 3 (3)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (13) | 7 (21) | 3 (3) | 3 (3) | 4 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (9) | 4 (4) | 4 (13) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (10) | 2 (3) | 1 (1) | 0 (0) | 2 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (5) | 0 (0) | 3 (14)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 5 (13) | 2 (6) | 1 (3) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenoviral upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmetria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary sediment abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cluster headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Central venous catheter removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of control of legs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04420598/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT04420598/SAP_001.pdf